CLINICAL TRIAL: NCT00393718
Title: Effect of Liraglutide on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1700
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Glyburide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide 0.9 mg + glibenclamide placebo
  Interventions: Drug: liraglutide; Drug: placebo
- Glibenclamide (Active Comparator): Glibenclamide 1.25-2.5 mg + liraglutide placebo
  Interventions: Drug: glibenclamide; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 0.9 mg/day. Injected s.c. (under the skin) once daily.
  Arms: Liraglutide
Drug: glibenclamide — 1.25-2.5 mg tablet. Given orally once or twice daily.
  Arms: Glibenclamide
Drug: placebo — liraglutide placebo. Injected s.c. (under the skin) once daily.
  Arms: Glibenclamide
Drug: placebo — glibenclamide placebo. Given orally once or twice daily.
  Arms: Liraglutide

SUMMARY:
This trial is conducted in Japan. The trial aims for comparison of the effect on glycaemic control of liraglutide, compared to sulfonylurea (SU treatment), as assessed by HbA1c after 24 and 52 weeks in subjects with type 2 diabetes. Trial has a randomisation period of 24 weeks followed by a 28 week extension period, in total 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diet/exercise therapy with or without an oral anti-diabetic drug for at least eight weeks
* HbA1c greater than or equal to 7.0% and less than 10.0%
* BMI (Body Mass Index) less than 35 kg/m2

Exclusion Criteria:

* Treatment with insulin within the last 12 weeks
* Treatment with any drug that could interfere with the glucose level
* Any serious medical condition
* Females who are pregnant, have intention of becoming pregnant or are breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Seino Y, Rasmussen MF, Nishida T, Kaku K. Efficacy and safety of the once-daily human GLP-1 analogue, liraglutide, vs glibenclamide monotherapy in Japanese patients with type 2 diabetes. Curr Med Res Opin. 2010 May;26(5):1013-22. doi: 10.1185/03007991003672551. PMID 20199137
- [Result] Seino Y, Rasmussen MF, Clauson P, Kaku K. The once-daily human glucagon-like peptide-1 analog, liraglutide, improves beta-cell function in Japanese patients with type 2 diabetes. J Diabetes Investig. 2012 Aug 20;3(4):388-95. doi: 10.1111/j.2040-1124.2012.00193.x. PMID 24843595
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Derived] Hegedus L, Moses AC, Zdravkovic M, Le Thi T, Daniels GH. GLP-1 and calcitonin concentration in humans: lack of evidence of calcitonin release from sequential screening in over 5000 subjects with type 2 diabetes or nondiabetic obese subjects treated with the human GLP-1 analog, liraglutide. J Clin Endocrinol Metab. 2011 Mar;96(3):853-60. doi: 10.1210/jc.2010-2318. Epub 2011 Jan 5. PMID 21209033
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 sites in Japan.
Pre-assignment Details: Subjects included in the study were patients with type 2 diabetes treated with diet therapy only or diet therapy and one OAD (Oral Anti-Diabetic Drug). Subjects on OAD therapy discontinued their current treatment during the run-in period (Weeks 4-6 before dosing). A total of 411 subjects were randomised, 11 subjects were not exposed to study drug.
Period: Overall Study
Arm/Group | Liraglutide | Glibenclamide
Started | 268 | 132
Completed | 225 | 110
Not Completed | 43 | 22
Not completed — Adverse Event | 20 | 8
Not completed — Protocol Violation | 1 | 2
Not completed — Lack of Efficacy | 10 | 9
Not completed — Hypoglycaemia | 3 | 2
Not completed — Subject decision | 5 | 0
Not completed — Withdrawal of consent | 2 | 1
Not completed — Missed measurement | 1 | 0
Not completed — Move | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Glibenclamide | Total
Number analyzed (Participants) | 268 | 132 | 400
Age, Customized [Number; unit: participants]
  20-29 years | 4 | 0 | 4
  30-39 years | 11 | 6 | 17
  40-49 years | 43 | 20 | 63
  50-59 years | 77 | 46 | 123
  60-69 years | 98 | 40 | 138
  70- years | 35 | 20 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.4) | 58.5 (10.4) | 58.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 46 | 131
  Male | 183 | 86 | 269
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 24.90 (3.69) | 24.62 (3.84) | 24.81 (3.74)
Body Weight [Mean (Standard Deviation); unit: kg] | 66.19 (12.61) | 65.43 (12.89) | 65.94 (12.69)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of diabetes
  years | 8.13 (6.68) | 8.48 (6.84) | 8.25 (6.73)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated Haemoglobin
  percentage of total haemoglobin | 8.27 (0.75) | 8.28 (0.78) | 8.28 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c) After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: Full Analysis Set (FAS) using LOCF (Last Observation Carried Forward) is all subjects who received at least one dose of study drug and have valid measurements both at baseline and at least one time point after baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 263 | 130
percentage of total haemoglobin | 6.99 (0.07) | 7.50 (0.09)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; ANOVA model included HbA1C at baseline as a covariate and treatment group and pre-trial treatment as fixed effects. Hypothesis for non-inferiority: H0: μ0.9 - μG ≥ 0.4, H1: μ0.9 - μG < 0.4, Hypothesis for superiority: H0: μ0.9 - μG ≥ 0.0, H1: μ0.9 - μG < 0.0, where μ0.9 and μG are population mean after 24-week treatment for liraglutide 0.9 mg/day and glibenclamide, respectively. When non-inferiority was confirmed, superiority was evaluated based on the closed testing procedure; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion: Upper limit of confidence interval of mean difference(= Liraglutide - Glibenclamide) is less than 0.4%. Superiority criterion: Upper limit of confidence interval of mean difference(= Liraglutide - Glibenclamide) is less than 0.0%; p < 0.0001, ANOVA — p-value is for the null hypothesis for superiority. A significance level of a one-sided 2.5% was used for statistical hypothesis testing; Least Squares Mean = -0.50, 95% CI [-0.70 to -0.30]

2. Secondary Outcome: Glycosylated Haemoglobin A1c (HbA1c) After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 263 | 130
percentage of total haemoglobin | 7.31 (0.08) | 7.80 (0.10)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; 95% confidence interval for the mean difference (liraglutide - glibenclamide) was calculated under an ANOVA model with treatment group and pre-trial treatment as fixed effects and corresponding baseline value as a covariate, and no statistical testing was performed; Test type: Superiority or Other; ANOVA; Least Squares Mean = -0.49, 95% CI [-0.71 to -0.27]

3. Secondary Outcome: Fasting Plasma Glucose After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 261 | 130
mg/dL | 137.2 (1.9) | 150.1 (2.5)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; The analysis was performed based on an ANOVA model with treatment group and pre-trial treatment as fixed effects and corresponding baseline value as a covariate. The following null hypothesis (H0) was statistically tested against the alternative hypothesis (H1). H0: μ0.9 = μG, H1: μ0.9 ≠ μG where μ0.9 and μG are population mean after 24-week treatment for liraglutide 0.9 mg/day and glibenclamide, respectively; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -12.9, 95% CI [-18.2 to -7.5]

4. Secondary Outcome: Fasting Plasma Glucose After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 261 | 130
mg/dL | 145.8 (2.4) | 157.5 (3.2)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -11.7, 95% CI [-18.6 to -4.9]

5. Secondary Outcome: Postprandial Glucose AUC After 24 Weeks of Treatment
Description: Postprandial glucose AUC measured 0-3 hours after a meal after 24 weeks of treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL *h
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 243 | 119
mg/dL *h | 557.54 (9.53) | 670.60 (12.69)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -93.05, 95% CI [-119.61 to -66.50]

6. Secondary Outcome: Postprandial Glucose AUC After 52 Weeks of Treatment
Description: Postprandial glucose AUC measured 0-3 hours after a meal after 52 weeks of treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL *h
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 228 | 112
mg/dL *h | 608.66 (11.18) | 683.17 (14.96)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -74.51, 95% CI [-105.75 to -43.27]

7. Secondary Outcome: Mean PG in 7-point Plasma Glucose Profile After 24 Weeks of Treatment
Description: Plasma glucose (PG) profile measured after 24 weeks of treatment. The time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 237 | 120
mg/dL | 155.98 (2.61) | 173.61 (3.51)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -17.63, 95% CI [-25.00 to -10.27]

8. Secondary Outcome: Mean PG in 7-point Plasma Glucose Profile After 52 Weeks of Treatment
Description: Mean plasma glucose(PG) in 7-point plasma glucose profile measured after 52 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 237 | 119
mg/dL | 167.39 (3.22) | 184.60 (4.34)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -17.21, 95% CI [-26.32 to -8.09]

9. Secondary Outcome: Mean Postprandial PG Increment in 7-point Plasma Glucose Profile After 24 Weeks of Treatment
Description: Mean postprandial plasma glucose (PG) increment in 7-point plasma glucose profile, ie the mean of the difference of plasma glucose measured before and after a meal, after 24 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 238 | 120
mg/dL | 59.69 (2.83) | 79.66 (3.75)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -19.97, 95% CI [-27.99 to -11.94]

10. Secondary Outcome: Mean Postprandial PG Increment in 7-point Plasma Glucose Profile After 52 Weeks of Treatment
Description: Mean postprandial plasma glucose (PG) increment in 7-point plasma glucose profile, ie the mean of the difference of plasma glucose measured before and after a meal, after 52 weeks of treatment. The 7 time points during the day were: Before breakfast, 120 minutes after start of breakfast, before lunch, 120 minutes after start of lunch, before dinner, 120 minutes after start of dinner, and at bedtime.
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 238 | 119
mg/dL | 63.56 (2.96) | 76.59 (3.94)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -13.03, 95% CI [-21.46 to -4.60]

11. Secondary Outcome: Body Weight After 24 Weeks of Treatment
Time Frame: after 24 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 265 | 130
kg | 64.06 (0.15) | 65.97 (0.20)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — A significance level of a two-sided 5% was used for statistical hypothesis testing; Least Squares Mean = -1.91, 95% CI [-2.34 to -1.48]

12. Secondary Outcome: Body Weight After 52 Weeks of Treatment
Time Frame: after 52 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 265 | 130
kg | 64.30 (0.19) | 66.01 (0.25)
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; ANOVA; Least Squares Mean = -1.71, 95% CI [-2.25 to -1.18]

13. Secondary Outcome: Hypoglycaemic Episodes
Description: Hypoglycaemic episodes measured over 52 weeks of treatment. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: over 52 weeks of treatment
Population: Full Analysis Set (FAS) consists of all subjects who received at least one dose of study drug.
Measure: Number; unit: number of events per year of exposure
Arm/Group | Liraglutide | Glibenclamide
Number analyzed (Participants) | 268 | 132
number of events per year of exposure
  All hypoglycaemic episodes | 0.694 | 3.843
  Major | 0.000 | 0.000
  Minor | 0.187 | 1.103
  Symptoms only | 0.507 | 2.740
Statistical Analysis 1: Comparison: Liraglutide vs Glibenclamide; The relative risk for 'All hypoglycaemic episodes' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 0.20, 95% CI [0.12 to 0.35]
Statistical Analysis 2: Comparison: Liraglutide vs Glibenclamide; The relative risk for 'Minor episodes' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 0.18, 95% CI [0.09 to 0.36]
Statistical Analysis 3: Comparison: Liraglutide vs Glibenclamide; The relative risk for 'Symptoms only' and 95% confidence interval are based on a generalised linear negative-binomial model, which included treatment group as a fixed effect and log of exposure time as an offset variable; Test type: Superiority or Other; Negative binomial regression model; Rate ratio = 0.20, 95% CI [0.11 to 0.34]

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time span over 52 weeks.
Description: The safety analysis population consists of all subjects exposed to study drug (Full Analysis Set, FAS).
Arm/Group | Liraglutide | Glibenclamide
Serious Adverse Events (participants affected / at risk) | 20/268 | 14/132
Other Adverse Events (participants affected / at risk) | 172/268 | 91/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=268) | Glibenclamide (N=132)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase MB (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=268) | Glibenclamide (N=132)
Nasopharyngitis (Infections and infestations) | 100 (183) | 57 (94)
Bronchitis (Infections and infestations) | 11 (13) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 26 (31) | 9 (12)
Constipation (Gastrointestinal disorders) | 21 (23) | 7 (8)
Stomach discomfort (Gastrointestinal disorders) | 14 (21) | 3 (5)
Nausea (Gastrointestinal disorders) | 14 (24) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 11 (11)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 25 (48) | 9 (10)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Diabetic retinopathy (Eye disorders) | 16 (16) | 9 (10)
Headache (Nervous system disorders) | 15 (22) | 6 (11)
Hypertension (Vascular disorders) | 11 (11) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.